CLINICAL TRIAL: NCT04163159
Title: Genetic Markers of Circulating Tumor DNA for Monitoring Breast Cancer in Patients of the Hospital San Juan de Dios From 2018 to 2020.
Brief Title: Genetic Markers of Circulating Tumor DNA for Monitoring Breast Cancer Patients in Costa Rica
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universidad de Costa Rica (Other)
Responsible Party: Sponsor
Other Study IDs: R018-SABI-00193; B9316 (Other: Universidad de Costa Rica)
Record Dates: First submitted 2019-11-06; First posted 2019-11-14 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Metastatic Breast Cancer; Mutation, Point
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and whole blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The use of circulating tumor DNA (ctDNA) as a noninvasive test for breast cancer monitoring throughout the course of the disease

DETAILED DESCRIPTION:
The concentrations of the cell free DNA (cfDNA) and somatic mutations in circulating tumor DNA (ctDNA) in serial samples correlate with the number of days of the progression-free period and with the overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic breast cancer before the start of chemotherapeutic treatment

Exclusion Criteria:

* Patients with incomplete clinical records

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Metastasic breast cancer females
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2019-01-07 (Actual); Primary Completion 2020-10-31 (Estimated); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
Assessment of circulating free DNA (cfDNA) concentration (in ng/uL) obtained from peripheral blood (liquid biopsy). | 12 months
  Samples will be analyze with Real time PCR and fluorometric assay and compare with overall survival
Number of somatic mutation findings in circulating free DNA (cfDNA) obtained from peripheral blood (liquid biopsy) | 12 months
  Samples will be analyze with targeted NGS sequencing panel

SECONDARY OUTCOMES:
Estrogen Receptor (ER), Progesterone Receptor (PR), Human Epidermal Growth Factor Receptor 2 (HER2) status | 24 months
  ER, PR, HER2 status
Overall survival of participant | 24 months
  Overall survival of participant
Cancer stage of participant | 24 months
  Cancer stage of participant

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital San Juan de Dios, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cristofanilli M, Budd GT, Ellis MJ, Stopeck A, Matera J, Miller MC, Reuben JM, Doyle GV, Allard WJ, Terstappen LW, Hayes DF. Circulating tumor cells, disease progression, and survival in metastatic breast cancer. N Engl J Med. 2004 Aug 19;351(8):781-91. doi: 10.1056/NEJMoa040766. PMID 15317891
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] Diaz LA Jr, Bardelli A. Liquid biopsies: genotyping circulating tumor DNA. J Clin Oncol. 2014 Feb 20;32(6):579-86. doi: 10.1200/JCO.2012.45.2011. Epub 2014 Jan 21. PMID 24449238
- [Background] Garcia-Saenz JA, Ayllon P, Laig M, Acosta-Eyzaguirre D, Garcia-Esquinas M, Montes M, Sanz J, Barquin M, Moreno F, Garcia-Barberan V, Diaz-Rubio E, Caldes T, Romero A. Tumor burden monitoring using cell-free tumor DNA could be limited by tumor heterogeneity in advanced breast cancer and should be evaluated together with radiographic imaging. BMC Cancer. 2017 Mar 22;17(1):210. doi: 10.1186/s12885-017-3185-9. PMID 28330468
- [Background] Goss PE, Lee BL, Badovinac-Crnjevic T, Strasser-Weippl K, Chavarri-Guerra Y, St Louis J, Villarreal-Garza C, Unger-Saldana K, Ferreyra M, Debiasi M, Liedke PE, Touya D, Werutsky G, Higgins M, Fan L, Vasconcelos C, Cazap E, Vallejos C, Mohar A, Knaul F, Arreola H, Batura R, Luciani S, Sullivan R, Finkelstein D, Simon S, Barrios C, Kightlinger R, Gelrud A, Bychkovsky V, Lopes G, Stefani S, Blaya M, Souza FH, Santos FS, Kaemmerer A, de Azambuja E, Zorilla AF, Murillo R, Jeronimo J, Tsu V, Carvalho A, Gil CF, Sternberg C, Duenas-Gonzalez A, Sgroi D, Cuello M, Fresco R, Reis RM, Masera G, Gabus R, Ribeiro R, Knust R, Ismael G, Rosenblatt E, Roth B, Villa L, Solares AL, Leon MX, Torres-Vigil I, Covarrubias-Gomez A, Hernandez A, Bertolino M, Schwartsmann G, Santillana S, Esteva F, Fein L, Mano M, Gomez H, Hurlbert M, Durstine A, Azenha G. Planning cancer control in Latin America and the Caribbean. Lancet Oncol. 2013 Apr;14(5):391-436. doi: 10.1016/S1470-2045(13)70048-2. PMID 23628188
- [Background] Overman MJ, Modak J, Kopetz S, Murthy R, Yao JC, Hicks ME, Abbruzzese JL, Tam AL. Use of research biopsies in clinical trials: are risks and benefits adequately discussed? J Clin Oncol. 2013 Jan 1;31(1):17-22. doi: 10.1200/JCO.2012.43.1718. Epub 2012 Nov 5. PMID 23129736
- [Background] PDQ Cancer Genetics Editorial Board. Genetics of Breast and Gynecologic Cancers (PDQ(R)): Health Professional Version. 2025 Mar 6. In: PDQ Cancer Information Summaries [Internet]. Bethesda (MD): National Cancer Institute (US); 2002-. Available from http://www.ncbi.nlm.nih.gov/books/NBK65767/ PMID 26389210
- [Background] Uehiro N, Sato F, Pu F, Tanaka S, Kawashima M, Kawaguchi K, Sugimoto M, Saji S, Toi M. Circulating cell-free DNA-based epigenetic assay can detect early breast cancer. Breast Cancer Res. 2016 Dec 19;18(1):129. doi: 10.1186/s13058-016-0788-z. PMID 27993161
- [Background] Yanagawa T, Kagara N, Miyake T, Tanei T, Naoi Y, Shimoda M, Shimazu K, Kim SJ, Noguchi S. Detection of ESR1 mutations in plasma and tumors from metastatic breast cancer patients using next-generation sequencing. Breast Cancer Res Treat. 2017 Jun;163(2):231-240. doi: 10.1007/s10549-017-4190-z. Epub 2017 Mar 10. PMID 28283903
- [Background] Ye Q, Qi F, Bian L, Zhang SH, Wang T, Jiang ZF. Circulating-free DNA Mutation Associated with Response of Targeted Therapy in Human Epidermal Growth Factor Receptor 2-positive Metastatic Breast Cancer. Chin Med J (Engl). 2017 Mar 5;130(5):522-529. doi: 10.4103/0366-6999.200542. PMID 28229982